CLINICAL TRIAL: NCT05295355
Title: Effect of Tiotropium Bromide Combined With Odaterol on Small Airway Remodeling in Patients With Mild to Moderate Chronic Obstructive Pulmonary Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Principal Investigator, ShiYue Li, Ph.D, Guangzhou Institute of Respiratory Disease
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: OCT-COPD
Record Dates: First submitted 2021-12-10; First posted 2022-03-25 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tiotropium Bromide Combined With Odaterol (Experimental): Tiotropium O Datlow inhalation spray 60 bottles per bottle, each containing 2.5 tiotropium ammonium g (equivalent to 3.124 g of thiotropium bromide) and 2.5 2.5 g (equivalent to 2.736 2.736 g of hydrochloric acid) by O Datlow. ® The inhaler was inhaled and administered twice a time, once a day, at the same time every day for 52 weeks
  Interventions: Drug: Tiotropium Bromide Combined With Odaterol
- Tiotropium Bromide (Experimental): Tiotropium Bromide Spray (Si Lihua ® Neng Beile ®）： 0.22624mg/ml (calculated by tiotropium), 60 strokes per bottle, containing 2.5 µ g of tiotropium bromide per stroke, through Neng Beile ® Inhaler inhalation administration, 2 presses per inhalation, once a day, administered at the same time every day for 52 weeks.
  Interventions: Drug: Tiotropium Bromide Combined With Odaterol

INTERVENTIONS:
Drug: Tiotropium Bromide Combined With Odaterol — 2 puffs once daily at the same time of the day for 52 week
  Other Names: Tiotropium BromideInhalation Aerosol Suspension

SUMMARY:
72 patients with mild to moderate chronic obstructive pulmonary disease were planned to be enrolled in this study and then treated with olodaterol combined with thiotropium bromide, and thiotropium bromide, respectively, for 52 weeks. To assess the effect of the test drug on small airway remodeling in patients.

DETAILED DESCRIPTION:
Studies have confirmed that thiotropium bromide combined with olodaterol can significantly improve airway inflammation, quality of life and pulmonary function in patients with stable COPD, without significantly increasing adverse reactions, which is worthy of clinical promotion. At present, there are few reports on the effect of thiotropium combined with olodaterol on airway remodeling in COPD patients, so this randomized, double-blind, parallel-controlled, single-center clinical trial was designed to compare the long-term effects of thiotropium combined with olodaterol, and thiotropium on small airway remodeling in patients with mild to moderate chronic obstructive pulmonary disease.

72 patients with mild to moderate chronic obstructive pulmonary disease were planned to be enrolled in this study. After screening examination, eligible subjects were randomly assigned to the test group or the control group in a 1:1 ratio and received olodaterol combined with thiotropium bromide, and thiotropium bromide, respectively, for 52 weeks. The effect of the test drug on small airway remodeling was assessed at 12, 26, and 52 weeks after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged ≥ 40 years;
* Meet the diagnostic criteria of COPD, and GOLD grade I - II;
* FEV1/FVC < 70% and FEV1 ≥ 50% of the expected value after the use of bronchodilators;
* Patients must be able to complete all study-related steps, voluntarily participate in this study and sign the informed consen.

Exclusion Criteria:

* Patients with asthma, active tuberculosis, lung cancer, bronchiectasis, sarcoidosis, pulmonary fibrosis, pulmonary hypertension, pulmonary embolism, bronchiolitis obliterans, paradoxical bronchospasm;
* Patients with blood eosinophilia;
* Patients with upper respiratory tract infection;
* Patients with liver or renal insufficiency;
* Patients with severe unstable systemic diseases or malignant tumors;
* Patients with glaucoma, benign prostatic hyperplasia or bladder neck obstruction;
* Patients with hypokalemia, hyperglycemia, diabetes, ketoacidosis or other serious systemic diseases such as heart, brain, liver, kidney, digestive system, endocrine system, immune system, blood;
* Women of childbearing age who are pregnant, lactating or plan to become pregnant;
* Patients who have undergone previous pneumonectomy or received lung volume reduction surgery within 12 months before screening;
* Patients with mental illness;
* Patients who have participated in other clinical trials within 3 months before screening;
* Allergic constitution or known allergy to atropine or its derivatives (such as isopropylamine or oxytoluium) Or those who are allergic to the intervention drugs and their ingredients;
* The researchers believe that it is not appropriate to participate in this clinical trial.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2021-01-25 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Effect of Tiotropium Bromide Combined With Odaterol on endobronchial lumen area change | at week 52
  difference in change from baseline in grade 7-9 endobronchial lumen area (Ai7-9) at week 52

SECONDARY OUTCOMES:
Effect of Tiotropium Bromide Combined With Odaterol on mean bronchial diameter change | at week 52
  difference in change from baseline in grade 7-9 mean bronchial diameter (Dmean7-9) at week 52
Effect of Tiotropium Bromide Combined With Odaterol on bronchial airway wall area change | at week 52
  difference in change from baseline in grade 7-9 bronchial airway wall area (Aw and Aw% 7-9) at week 52
Effect of Tiotropium Bromide Combined With Odaterol on FEV1 change | at week 52
  difference in change from baseline in trough FEV1 at week 52
Effect of Tiotropium Bromide Combined With Odaterol on SGRQ total score change | at week 52
  difference in change from baseline in SGRQ （ST george's respiratory questionaire）total score at week 52
Effect of Tiotropium Bromide Combined With Odaterol on resonance frequency change | at week 52
  difference in change from baseline in resonance frequency (Fres) at week 52
Effect of Tiotropium Bromide Combined With Odaterol on peripheral airway resistance change | at week 52
  difference in change from baseline in peripheral airway resistance (R5-R20) at week 52
Effect of Tiotropium Bromide Combined With Odaterol on CAT total score change | at week 52
  difference in change from baseline in CAT（Chronic obstructive pulmonary disease assessment test） total score at week 52
Effect of Tiotropium Bromide Combined With Odaterol on mMRC total score change | at week 52
  difference in change from baseline in mMRC（Modified British medical research council） total score at week 52

CONTACTS AND LOCATIONS:
Overall Officials: Shiyue Li, Doctor, Principal Investigator — Guangzhou Institute of Respiratory Disease
Locations (1):
- Guangzhou Institute of Respiratory Diseases, Guangzhou, Guangdong, China